CLINICAL TRIAL: NCT00204958
Title: Evaluation of Glutamine Popsicles in Adult/Pediatric Bone Marrow Transplant (BMT)/Hematopoietic Stem Cell Transplant (HSCT) Patients
Brief Title: Glutamine Popsicles in Bone Marrow Transplant (BMT)/Hematopoietic Stem Cell Transplant (HSCT) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2003-222
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2015-10-01 (Estimated); Status verified 2015-09

CONDITIONS: Bone Marrow Transplantation; Hematopoietic Stem Cell Transplantion
Keywords: bone marrow transplant (BMT); hematopoietic stem cell transplant (HSCT)
MeSH Terms: interventions — Dietary Supplements

INTERVENTIONS:
Drug: nutritional supplement
Drug: glutamine popsicle

SUMMARY:
Nutrition is an important part of the recovery process after having a head injury so that subjects can gain strength and fight off infection. Liquid nutrition formulas are often given to patients through a tube that has been placed into the intestines for feeding when they are unable to eat on their own. Some reports suggest that nutrition with extra amounts of the amino acid called glutamine may decrease infections and hospital stay in severely injured patients. The purpose of this study is to evaluate if giving extra amounts of an amino acid called glutamine with liquid nutrition formulas will decrease the risk of infection and length of stay in the intensive care unit after having a head injury.

ELIGIBILITY:
Inclusion Criteria:

* Males
* Nonpregnant females
* Receiving chemotherapy for BMT/HSCT

Exclusion Criteria:

* Documented hepatic dysfunction
* History of cirrhosis
* History of acute renal failure (creatinine clearance < 25 mL/min)
* Gastrointestinal malabsorptive disorder

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2004-02; Primary Completion 2007-05 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
grade of mucositis

SECONDARY OUTCOMES:
need for intravenous versus oral nutritional supplementation

CONTACTS AND LOCATIONS:
Overall Officials: Gordon S Sacks, PharmD., FCCP, BCNSP, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States